CLINICAL TRIAL: NCT02555839
Title: Multicenter Non-interventional Study to Investigate Drug Utilization of Pomalidomide in Clinical Practice for the Treatment of Relapsed/Refractory Multiple Myeloma (rrMM)
Brief Title: Treatment of Relapsed/Refractory Multiple Myeloma (rrMM) With Pomalidomide in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-4047-MM-017
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma; Pomalidomide; Imnovid; Non-interventional
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone; dexamethasone acetate; Bortezomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pomalidomide and Dexamethasone: Pomalidomide 4mg capsules by mouth (PO) on days 1 through 21 of a 28 day cycle and Dexamethasone 40mg PO (≤75 years) or 20mg (>75years) on Days 1, 8, 15, 22 of a 28 day cycle until progression or unacceptable toxicity
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Pomalidomide, Bortezomib and Dexamethasone: Cycle 1-8: Pomalidomide 4mg capsules by mouth (PO) on days 1 through 14 of a 21 day cycle, Bortezomib (1,3mg/m2) s.c. on day 1, 4, 8, 11 of a 21 day cycle, and Dexamethasone 20mg PO (≤75 years) or 10mg (>75years) on Days 1, 2, 4, 5, 8, 9, 11, 12 of a 21 day cycle until progression or unacceptable toxicity; from cycle 9 onwards: Pomalidomide 4mg capsules by mouth (PO) on days 1 through 14 of a 21 day cycle, Bortezomib (1,3mg/m2) s.c. on day 1 and 8 of a 21 day cycle, and Dexamethasone 20mg PO (≤75 years) or 10mg (>75years) on Days 1, 2, 8, 9 of a 21 day cycle until progression or unacceptable toxicity
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Pomalidomide — 4mg capsule on d1 through 21 of a 28 day cycle
  Other Names: CC-4047; Imnovid
  Groups: Pomalidomide and Dexamethasone
Drug: Dexamethasone — 40 mg (≤75 years) or 20mg (>75 years) oral on d1, 8, 15, 22 of a 28 day cycle
  Other Names: Fortecortin
  Groups: Pomalidomide and Dexamethasone
Drug: Pomalidomide — 4mg capsule on d1 through 14 of a 21 day cycle
  Groups: Pomalidomide, Bortezomib and Dexamethasone
Drug: Dexamethasone — cycle 1-8: 20mg PO (≤75 years) or 10mg (>75years) on Days 1, 2, 4, 5, 8, 9, 11, 12 of a 21 day cycle; from cycle 9 onwards: Dexamethasone 20mg PO (≤75 years) or 10mg (>75years) on Days 1, 2, 8, 9 of a 21 day cycle
  Groups: Pomalidomide, Bortezomib and Dexamethasone
Drug: Bortezomib — cycle 1-8: Bortezomib (1,3mg/m2) s.c. on day 1, 4, 8, 11 of a 21 day cycle; from cycle 9 onwards: Bortezomib (1,3mg/m2) s.c. on day 1 and 8 of a 21 day cycle,
  Groups: Pomalidomide, Bortezomib and Dexamethasone

SUMMARY:
There is a high unmet medical need for an anti-myeloma therapy for RRMM patients previously treated with Lenalidomide and Bortezomib, due to poor prognosis.

This observational study focuses on the collection of data concerning the safe and optimal usage of Pomalidomide, a new therapy option for RRMM patients, thereby increasing the knowledge about optimal AE management. Beside this, further analysis of tolerability, dosage and efficacy will be performed.

This knowledge could lead to a optimization of Pomalidomide usage and treatment.

DETAILED DESCRIPTION:
There is a high unmet medical need for further anti-myeloma therapy in patients with RRMM who have previously been treated with Lenalidomide and Bortezomib containing regimens that is both active and tolerable, as these patients have a poor prognosis. Hands-on experience with Pomalidomide is very limited in Austria and a non-interventional study enhances the attention paid to safe use and handling of the product as well as increase knowledge about optimal adverse event (AE) management substantially.

A detailed record of the medical history including. co-morbidities and pre-treatment regimens will allow analysis of the impact there of on tolerability, dosage and efficacy.

Beside the collection of data on efficacy and tolerability this observational drug utilization study could give insight into the clinical practice and the routine use of Pomalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Signed IC
* age ≥ 18 years
* relapsed/refractory MM
* cohort A (combination pomalidomide und dexamethasone):

  ≥2 antimyeloma treatments (including lenalidomide and bortezomib), induction therapy followed by ASCT and consolidation or maintenance therapy is considered as 1 antimyeloma treatment
* cohort B (combination pomalidomide, bortezomib and dexamethasone):

  ≥1 antimyeloma treatments (including lenalidomide) induction therapy followed by ASCT and consolidation or maintenance therapy is considered as 1 antimyeloma treatment
* refractory to last antimyeloma treatment
* adequate contraception according to RMP
* adequate thrombosis prophylaxis

Exclusion Criteria:

1. Pregnant or Lactating Females
2. Known hypersensitivity to Imnovid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed and/or Refractory Multiple Myeloma
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Up to 2 years
  The number of participant adverse events

SECONDARY OUTCOMES:
Response Rate | Up to 2 years
  The number of participants who achieve a response
Progression Free Survival | Up to 2 years
  The number of participants who survive without progression of disease
Duration of Response | Up to 2 years
  Duration of response is defined as time from the initial documented response (partial response or better) to confirmed disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- Austria (13):
  - LKH Feldkirch, Intern E, Hämatologie, Feldkirch
  - Medical University Graz, Graz
  - KH der Elisabethinen Linz , 1. Interne Hämato-Onkologie, Linz
  - Kepleruniversitätsklinikum GmbH, Hämatologie und Internistische Onkologie, Linz
  - Krankenhaus der Barmherzigen Schwestern Ried, Innere Medizin I, Ried
  - SCRI-CCCIT gemeinnützige GmbH & Universitätsklinikum der PMU Salzburg Gemeinnützige Salzburger Landeskliniken BetriebsgmbH, Salzburg
  - LKH Steyr, Innere Medizin II, Steyr
  - AKH, Innere Medizin I, Klin. Abt. f. Hämatologie, Vienna
  - AKH, Universitätsklinik für Innere Medizin I /Klin. Abteilung für Onkologie, Vienna
  - St. Josef Krankenhaus Wien,1. Abteilung für Innere Medizin Zentrum für Onkologie, Vienna
  - Hanusch Krankenhaus Wien 3. Medizinische Abteilung Hämatolog, Vienna
  - Wilhelminenspital, 1. Med.Abteilung, Zentrum für Onkologie, Vienna
  - Salzkammergut-Klinikum Vöcklabruck, Abteilung Innere Medizin, Vöcklabruck

REFERENCES:
- See also: Expanded Access for CC-4047 — https://clinicaltrials.gov/ct2/show/NCT03723096?term=NCT03723096&rank=1